CLINICAL TRIAL: NCT06460376
Title: Comparative Effects of Wurn Technique and Mercier Therapy on Dyspareunia, Dysmenorrhea, and Quality of Life in Women With Endometriosis
Brief Title: Comparative Effects of Wurn Technique and Mercier Therapy in Women With Endometriosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0563
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Endometriosis
Keywords: Dyspareunia; Dysmenorrhea; endometriosis
MeSH Terms: conditions — Endometriosis; Dyspareunia; Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wurn technique (Experimental): The principle intent of the Wurn Technique is to decrease pain and increase mobility and function of abdominopelvic and reproductive organs by diminishing adhesions. The protocol focuses on deforming the adhesive collagen cross-links comprising adhesions that appear to contribute to the underlying causes of endometriosis.
  Interventions: Other: Wurn Technique
- Mercier therapy (Active Comparator): The principal intent of mercier therapy is visceral pelvic manipulation that addresses scar tissue, adhesions, and the misalignment of pelvic organs. It increases blood flow and circulation to the pelvis.
  Interventions: Other: Mercier Therapy

INTERVENTIONS:
Other: Wurn Technique — Treatment:
  Site-specific pressures for 30 seconds across the restrictive bands of adhered tissues and structures, working progressively deeper from the most superficial tissues Traction: focusing on these adhered areas, engage the uterine fundus and sidewalls and traction them to the left.
  To assist and improve the mobility of the soft tissues, release the traction tension either suddenly or gradually, depending on the desired effect to decrease spasms and adhesions between the uterus and the bladder. The baseline treatment was moist heat.
  Each therapy session was 30 minutes for 6 weeks and 2 sessions per week. 10 minutes for baseline treatment.
  Arms: Wurn technique
Other: Mercier Therapy — Treatment:
  The patient lay face up on a massage or exam table. Feel viscera, major internal organs located in the abdomen by lightly pressing through abdominal muscles.
  Manual poking, pressing, and massage actions do three things:
  Reveals visceral adhesions. Find tender spots. Breaks up adhesions. Massaging and pressing stretch the collagen fibers that make up fascia, which loosens tightly bound fibers to break up adhesions. This releases the organs and allows them to move more freely.
  Abdominal massage with pressing, deep strokes, and friction. The baseline treatment was moist heat. Each therapy session was 25 minutes for 6 weeks and 1 session per week. 10 minutes for baseline treatment
  Arms: Mercier therapy

SUMMARY:
This project was a Randomized controlled trial conducted to check the comparative effects of wurn technique and mercier therapy on dyspareunia, dysmenorrhea, and quality of life in women with endometriosis. The duration was 6 months, convenient sampling was done, subjects following eligibility criteria from DHQ Hospital Narowal and THQ Hospital Shakargarh were randomly assigned, a baseline assessment was done, Group A participants were given baseline treatment along with wurn technique 2 sessions per week for 6 weeks, Group B participants were given baseline treatment along with mercier therapy 1 session per week for 6 weeks, the post-intervention assessment was done, via the Marinoff Scale, Mankoski Pain Scale and Endometriosis Health Profile Questionnaire (EHP 30). Data was analyzed by using SPSS version 26.

Detailed Description: Endometriosis

DETAILED DESCRIPTION:
Endometriosis is the condition involving the presence of glands or stroma of the endometrial lining outside the uterus cavity. Its characteristics include unpleasant pain in the pelvic region, impaired fertility, pain during or after sex, and heavy bleeding during periods. Endometriosis occurs as a result of genetic, angiogenic, immunological, and inflammatory factors. In endometriosis, adhesions may be formed due to local inflammation. It can also occur as the blood-filled implants start bleeding in their surroundings. As a result of this bleeding healing occurs which causes scar formation. Pharmacologically, NSAIDS are used for instant pain relief. The most common surgical approach is laparoscopy. Physiotherapy in its various forms can be an excellent complement to the gynecological treatment of endometriosis. as previous studies also reported the effect of pelvic massage, pelvic manipulation, kinesiotherapy, and hydrotherapy. According to researcher knowledge, there is limited evidence on wurn technique and mercier therapy and how these techniques improve dyspareunia, dysmenorrhea, and quality of life in women with endometriosis. This study aims to see the comparative effects of wurn technique and mercier therapy on dyspareunia, dysmenorrhea, and quality of life in women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 25-43(17)
* Diagnosed patients with endometriosis
* BMI (18.5-29.9),(normal and overweight)
* Multigravida
* Mode of delivery: vaginal delivery or c section both
* Females having grade 1 or 2 grade on the dyspareunia scale
* Females having moderate scores on EHP -30

Exclusion Criteria:

* Malignancy
* Pregnancy
* Fibroids
* Pelvic congestion syndrome
* Pelvic inflammatory disease
* Females having IUD (inter uterine device)
* Recent abdominal or pelvic surgery
* Ovarian abscess

Ages: 25 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Endometriosis Health Profile Questionnaire (EHP 30) | 6 Weeks
  Endometriosis health profile questionnaire (EHP 30) is to evaluate the suitably self- report health status. It involves 30 items to identify the health status of patients with endometriosis.A core questionnaire which consists of five scales (pain, control and powerlessness, emotional well-being support and self-image). Internal consistency reliability is high for all dimensions (alpha ranged from 0.84 to 0.91)

SECONDARY OUTCOMES:
Mankoski Pain Scale | 6 weeks
  The Mankoski Pain Scale is a numerical scale ranging from zero to 10: zero indicates no pain and 10 represents pain so severe that an individual loses consciousness. It will be used to indicate dysmenorrhea.The reliability of mankoski scale is 0.84

OTHER OUTCOMES:
Marinoff Scale | 6 weeks
  Marinoff scale is used to evaluate dyspareunia. It includes 4 choices with a score of 0-3. Reliability of the scale was obtained with a Cronbach's alpha of 0.94

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - DHQ Hospital Narowal, Narowal, Punjab Province
  - THQ Hospital Shakargarh, Shakargarh, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koninckx PR, Fernandes R, Ussia A, Schindler L, Wattiez A, Al-Suwaidi S, Amro B, Al-Maamari B, Hakim Z, Tahlak M. Pathogenesis Based Diagnosis and Treatment of Endometriosis. Front Endocrinol (Lausanne). 2021 Nov 25;12:745548. doi: 10.3389/fendo.2021.745548. eCollection 2021. PMID 34899597
- [Background] Lee SY, Koo YJ, Lee DH. Classification of endometriosis. Yeungnam Univ J Med. 2021 Jan;38(1):10-18. doi: 10.12701/yujm.2020.00444. Epub 2020 Aug 7. PMID 32764213
- [Background] International Working Group of AAGL, ESGE, ESHRE and WES; Tomassetti C, Johnson NP, Petrozza J, Abrao MS, Einarsson JI, Horne AW, Lee TTM, Missmer S, Vermeulen N, Zondervan KT, Grimbizis G, De Wilde RL. An international terminology for endometriosis, 2021. Hum Reprod Open. 2021 Oct 22;2021(4):hoab029. doi: 10.1093/hropen/hoab029. eCollection 2021. PMID 34693033
- [Background] Vallve-Juanico J, Houshdaran S, Giudice LC. The endometrial immune environment of women with endometriosis. Hum Reprod Update. 2019 Sep 11;25(5):564-591. doi: 10.1093/humupd/dmz018. PMID 31424502
- [Background] Smolarz B, Szyllo K, Romanowicz H. Endometriosis: Epidemiology, Classification, Pathogenesis, Treatment and Genetics (Review of Literature). Int J Mol Sci. 2021 Sep 29;22(19):10554. doi: 10.3390/ijms221910554. PMID 34638893
- [Background] Kapoor R, Stratopoulou CA, Dolmans MM. Pathogenesis of Endometriosis: New Insights into Prospective Therapies. Int J Mol Sci. 2021 Oct 28;22(21):11700. doi: 10.3390/ijms222111700. PMID 34769130
- [Background] Arafah M, Rashid S, Akhtar M. Endometriosis: A Comprehensive Review. Adv Anat Pathol. 2021 Jan;28(1):30-43. doi: 10.1097/PAP.0000000000000288. PMID 33044230
- [Background] Christ JP, Yu O, Schulze-Rath R, Grafton J, Hansen K, Reed SD. Incidence, prevalence, and trends in endometriosis diagnosis: a United States population-based study from 2006 to 2015. Am J Obstet Gynecol. 2021 Nov;225(5):500.e1-500.e9. doi: 10.1016/j.ajog.2021.06.067. Epub 2021 Jun 17. PMID 34147493